CLINICAL TRIAL: NCT01838239
Title: Development of a Metabolic Assessment Tool for Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200715313
Record Dates: First submitted 2013-04-18; First posted 2013-04-24 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Immunoglobulin A Nephropathy; Healthy Subjects
Keywords: Fish oil; Omega-3 fatty acids
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Fish Oils

ARMS (1):
- Fish oil (Experimental)
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — Ocean Nutrition Fish Oil Capsules containing 1.9 g eicosapentaenoic acid (EPA) and 1.5 g docosahexaenoic acid (DHA)

SUMMARY:
The purpose of this study is to examine the variation between individuals in blood lipid metabolites, and the changes in these metabolites in response to omega-3 fatty acids in patients with immunoglobulin A nephropathy (IgAN) and in healthy subjects. The hypothesis is that measuring variation among individuals and changes in response to omega-3 fatty acids comprehensively by using metabolomics will help to identify those individuals who are responders and those who are non-responders to omega-3 fatty acids as an anti-inflammatory intervention.

DETAILED DESCRIPTION:
It is unclear how metabolomic profiles of individuals change in response to short-term intervention with omega-3 fatty acids. It is necessary to establish the means and standard deviations in the levels of omega-3 fatty acids and their related metabolites in healthy subjects and in different disease states in order to better understand the mechanisms related to lipid metabolism of metabolic diseases that are modified by omega-3 fatty acids. Specifically, the project will examine the metabolomic profiles of healthy controls and patients with immunoglobulin A nephropathy (IgAN) before and after an omega-3 fatty acid intervention. The IgAN patient samples were obtained from collaborators from a previously completed project. The healthy subjects were tested in a small pilot trial conducted at UC Davis as described below.

* Twelve healthy volunteers willing and able to take 6 g of fish oil for 6 weeks were recruited from the general UC Davis population including students, faculty, and staff. The volunteers were recruited by personal communication at seminars and other school-related activities as well as flyers posted on campus.
* The volunteers were contacted and scheduled for a screening and consent visit. Subjects who met all eligibility criteria and signed a consent form were then scheduled for a baseline blood draw and to collect a first morning urine sample. A research team member contacted each subject the day before their first scheduled study date to confirm and remind the subject about fasting, about collecting the first morning urine void, and the time and location of the study.
* On each study visit, the participants came to the Ragle Human Nutrition Center (1283 Academic Surge) between 7 and 9 am after an overnight fast, at which point they were weighed (clothed but with no shoes) on a digital scale and their height was measured. A registered phlebotomist drew 20 mL of blood by venipuncture for their baseline blood draw. Subjects also brought in their first morning urine sample at this time. Subjects were then given their fish oil capsules that were separated in a Ziploc bag for each week of the intervention. Subjects took the fish oil capsules at home at their own discretion but study personnel suggested they take the capsules after their last meal of the day and before bed each evening. Study personnel contacted subjects throughout the course of the study by phone and/or e-mail to make sure that there were no adverse effects from the fish oil and to ensure compliance. Subjects were instructed to record their diets through 24-hour dietary recalls before the baseline blood draw, and at 3 additional time points throughout the study.
* Immediately after blood collection, the researchers separated the red blood cells and peripheral blood mononuclear cells (PBMC) from the plasma, aliquoted the samples, and then stored them in a -70°C freezer for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* Weight at least 110 pounds or BMI at least 19
* Adult (aged 18-65 years old)
* Disclose which medications currently taking
* Able to come to the Ragle Center at the designated times
* Able to give blood
* Able to take 6 g fish oil per day for 6 weeks
* Able to carry out first morning urine collection
* Able to stop or avoid taking NSAIDS and allergy medications for 6 weeks
* Able to stop or avoid eating seafood and seaweed for 6 weeks

Exclusion Criteria:

* Pregnant or nursing (or unsure if pregnant)
* Diagnosed with a disease by their physician
* Currently taking prescription medications that alter lipid metabolism (such as HMG CoA reductase inhibitors, PPAR agonists, steroids) and/or anti-coagulants
* Currently has some form of anemia (or unsure)
* Has an existing health condition or concern
* Unable to stop or avoid taking NSAIDS and allergy medications for 6 weeks
* Unable to stop or avoid eating seafood or seaweed for 6 weeks
* Unable to give blood or do first morning urine collection
* Recently recovering from a major injury, infection, or illness (in the last 2-4 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Plasma lipid metabolomic profile | Baseline vs. 6 weeks
  Plasma lipid metabolomic profile includes fatty acids within lipid classes, oxylipins, lipoprotein particle size and distribution

SECONDARY OUTCOMES:
PBMC gene expression | Baseline vs. 6 weeks
  Measurement of changes in gene expression in peripheral blood mononuclear cells

OTHER OUTCOMES:
Urinary oxylipins | Baseline vs. 6 weeks
  Measurement of urinary oxylipins

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Hammock, PhD, Principal Investigator — University of California, Davis; Angela M Zivkovic, PhD, Principal Investigator — University of California, Davis; J. Bruce German, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Davis, California, United States

REFERENCES:
- [Derived] Berthelot CC, Kamita SG, Sacchi R, Yang J, Nording ML, Georgi K, Hegedus Karbowski C, German JB, Weiss RH, Hogg RJ, Hammock BD, Zivkovic AM. Changes in PTGS1 and ALOX12 Gene Expression in Peripheral Blood Mononuclear Cells Are Associated with Changes in Arachidonic Acid, Oxylipins, and Oxylipin/Fatty Acid Ratios in Response to Omega-3 Fatty Acid Supplementation. PLoS One. 2015 Dec 16;10(12):e0144996. doi: 10.1371/journal.pone.0144996. eCollection 2015. PMID 26672987